CLINICAL TRIAL: NCT06529445
Title: Food Effect and Relative Bioavailability Study of VC004 Capsules in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VC004-105
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-07

CONDITIONS: Locally Advanced or Metastatic Solid Tumor Harboring an NTRK Gene Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Dose VC004 group (Experimental)
  Interventions: Drug: High Dose VC004 Capsules
- Median Dose VC004 group (Experimental)
  Interventions: Drug: Median Dose VC004 Capsules
- Low Dose VC004 group (Experimental)
  Interventions: Drug: Low Dose VC004 Capsules

INTERVENTIONS:
Drug: High Dose VC004 Capsules — VC004 Capsules qd per period, for two periods
  Arms: High Dose VC004 group
Drug: Median Dose VC004 Capsules — VC004 Capsules qd per period, for two periods
  Arms: Median Dose VC004 group
Drug: Low Dose VC004 Capsules — VC004 Capsules qd per period, for two periods
  Arms: Low Dose VC004 group

SUMMARY:
This study will adopt a randomized, open-label, two-period, 2-way crossover design to evaluate Food effect and Relative bioavailability of VC004 Capsules in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent before study, and fully understand the study content, process and possible adverse reactions;
2. Able to complete the study in compliance with the protocol;
3. Subject (including partner) is willing to voluntarily take effective contraceptive measures from screening through 6 months after the last dose of study drug (see Appendix 5 for details);
4. Male and female subjects between the ages of 18 and 45 years, inclusive;
5. At least 50.0kg for male subjects, 45.0kg for female subjects, with a Body Mass Index (BMI= Weight/Height2) between 19.0-26.0 kg/m2, inclusive;

Exclusion Criteria:

1. More than 5 cigarettes per day on average within 3 months prior to screening;
2. with a history of allergies, including medication, food, mites, etc., or those known to be potentially allergic to drugs of the same class as the study drug;
3. History of drug and/or alcohol abuse (alcoholism defined as: drinking 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine); history of drug abuse or or have used drugs within the past five years;
4. Donation or loss of a significant volume of blood (> 400 mL) within 3 months prior to screening;
5. History of difficulties in swallowing or any history of gastrointestinal(such as reflux esophagitis, peptic ulcer, chronic diarrhea, chronic constipation), liver, kidney disease (whether cured or not) or surgery that affects drug absorption or excretion within 6 months prior to screening;
6. Those who Have taken strong inhibitors and / or inducers of liver metabolic enzymes (CYP1A2, 2A6, 2b6, 2c8, 2c19, 3A4 and 3A5) within 28 days prior to screening :strong inhibitors of liver metabolic enzymes such as ciprofloxacin, clopidogrel, itraconazole, ketoconazole, ritonavir, oleandomycin etc., strong inducers of liver metabolic enzymes such as rifampicin, carbamazepine, phenytoin sodium, St. John's wort, etc; Those who Have taken inhibitors and inducers of P-gp, MRPs, BCRP, OATP and other transporters and transporters within 28 days prior to screening; See Appendix 5 for details;
7. Intake of any prescription drugs, over-the-counter drugs, vitamin or herbal medicine within 14 days prior to screening;
8. Taking foods that affect CYP3A4 metabolism, such as grapefruit or drinks containing grapefruit within 2 weeks prior to screening, or taking high-intensity physical exercises (such as strength training, aerobic training and football playing) within 7 days prior to screening, or any other factors that affect drug absorption, distribution, metabolism and excretion;
9. Participated in other clinical trials within 3 months before screening (if the subject withdraws from the study before treatment, i.e. has not been randomized or received treatment, he or she can be enrolled in the study);
10. Those who cannot tolerate high-fat meals or have special requirements for diet and cannot accept unified diet；
11. A clinically significant vital signs abnormality during screening (body temperature (axillary temperature) < 36.0 ℃ or > 37.0 ℃; Pulse < 60bpm or > 100bpm; Systolic blood pressure <90mmhg or ≥ 140mmHg, diastolic blood pressure <60mmhg or ≥ 90mmHg);
12. A clinically significant 12-lead ECG abnormality;
13. Positive test results of blood pregnancy or is lactating for female subjects;
14. Any clinically significant abnormalities/findings in laboratory tests, or any clinically significant disease including but not limited to gastrointestinal, renal, hepatic, neurological system, blood, endocrine, tumor, lung, immune, mental, or cardiovascular and cerebrovascular diseases;
15. Positive test results for viral hepatitis (including hepatitis B and C), HIV antibody or syphilis antibody during screening;
16. Acute illness or concomitant medication from screening to the first dosing of study medication;
17. Consumption of chocolate or any food or beverages containing caffeine or (rich containing) xanthine within 24 h prior to screening;
18. Consumption of any product containing alcohol within 24 h prior to screening, or positive results from a screen for alcohol;
19. Positive results from a screen for urine drug test;
20. Cannot tolerate venipuncture and have a history of needle and blood sickness;
21. Subjects with Lactose intolerant;
22. Subjects were vaccinated within 4 weeks prior to screening, or planned to be vaccinated during the trial;
23. Any condition which in the opinion of Investigator is not suitable for subjects to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day1-Day7
Peak time(Tmax) | Day1-Day7
Area Under the Curve From Time Zero to Last Quantifiable Concentration(AUC） | Day1-Day7

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital,Affiliated to Southeast University, Nanjing, Jiangsu, China